CLINICAL TRIAL: NCT01460316
Title: Conotruncal Cardiac Defects and Metabolism, Nutrigenetic Factors of Etiopathogeny of Conotruncal Cardiac Defects
Brief Title: Conotruncal Cardiac Defects and Nutrigenetic Etiopathogeny
Acronym: CCOMET
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Universitaire Dijon (Other); CHU de Reims (Other)
Responsible Party: Principal Investigator, FEILLET François, Professor, M.D. Ph.D, Central Hospital, Nancy, France
Other Study IDs: 2011-A00346-35
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Conotruncal Cardiac Defects
Keywords: Conotruncal cardiac defects; methylation; genotype; cobalamin; folates; nutrition
MeSH Terms: conditions — Conotruncal cardiac defects | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Conotruncal cardiac defects patients
  Interventions: Biological: Bood sampling for biochemicals and genetic analysis
- Mothers of patients
  Interventions: Biological: Bood sampling for biochemicals and genetic analysis

INTERVENTIONS:
Biological: Bood sampling for biochemicals and genetic analysis — There will be one blood sampling for the nutritionnal, metabolic and genetic parameters studied in the protocol

SUMMARY:
The investigators planned to study the etiopathogenic factors of conotruncal cardiac defects regarding the relations between the metabolic, the genetic and the environmental factors which lead to these cardiopathy.

ELIGIBILITY:
Inclusion Criteria:

* Conotruncal cardiac defects patients and theirs mothers
* Weight: > 3750 g

Exclusion Criteria:

* Syndromic conotruncal cardiac defects
* 22q11 deletion Holder's
* Patients whose mother's took anti-folates before and during first pregnancy semester

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Conotruncal cardiac defects population and theirs mothers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François FEILLET, MD-PHD, Principal Investigator — CHU de Nancy- Hôpital Brabois Enfants
Locations (1):
- Service de Cardiologie Pédiatrique, CHU Brabois Enfants, Vandœuvre-lès-Nancy, France